CLINICAL TRIAL: NCT01981096
Title: Fibromyalgia Integrative Training for Teens
Acronym: FIT Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AR063412 (NIH); R21AR063412 (NIH)
Record Dates: First submitted 2013-10-24; First posted 2013-11-11 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Juvenile Fibromyalgia
Keywords: juvenile fibromyalgia; pain in children; musculoskeletal pain; cognitive behavioral therapy; coping skills training
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibromyalgia Integrative Training (Experimental): 8 week (16 sessions) combined intervention with cognitive-behavioral therapy and neuromuscular training
  Interventions: Behavioral: Fibromyalgia integrative training
- Cognitive Behavioral Therapy (Active Comparator): 8 week (16 session) cognitive-behavioral therapy treatment.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Fibromyalgia integrative training — Combined intervention with neuromuscular exercise training and cognitive behavioral therapy
  Arms: Fibromyalgia Integrative Training
Behavioral: Cognitive Behavioral Therapy — Therapy focused on training in behavioral pain coping skills
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this pilot randomized trial is to determine whether the fibromyalgia integrative training (FIT Teens) intervention is superior to cognitive-behavioral therapy (CBT) alone in reducing pain among adolescents with juvenile fibromyalgia (JFM).

Hypothesis 1: Patients in the FIT Teens group will show significantly greater reduction in pain intensity than the CBT group at final study assessment (i.e., 3-month follow up).

Hypothesis 2: Patients in both the FIT Teens and CBT groups will show significant reductions in functional disability and depressive symptoms at final study assessment (i.e., 3-month follow up).

DETAILED DESCRIPTION:
CBT has been found to have beneficial effects on improving coping among adolescents with JFM and increasing patients' ability to engage in daily activities. The purpose of this study is to evaluate whether CBT can be enhanced with specialized neuromuscular training, in the new fibromyalgia integrative training (FIT Teens) intervention, to produce stronger pain reduction than CBT alone. Neuromuscular training originates from the field of pediatric sports medicine and has been successfully used for injury prevention but has never before been utilized for pain management in JFM. This type of training emphasizes education and proper training in fundamental movement skills prior to the initiation of more vigorous physical activity and exercise. It is expected that the neuromuscular training integrated with established CBT techniques will enhance patients' ability to engage in exercise and to achieve better JFM pain control. Adolescents with JFM will be randomly assigned to receive either the 8-week FIT Teens intervention or an 8-week CBT program with assessments at baseline, post-treatment and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 12-18
* Juvenile fibromyalgia (JFM) diagnosed by a pediatric rheumatologist or pain physician using 2010 American College of Rheumatology (ACR) criteria and confirmation with a tender point exam of ≥ 11 of 18 tender points upon palpation
* Functional Disability Score ≥13 indicating at least moderate disability
* Average pain intensity in the past week ≥ 4 on a 0-10 cm Visual Analog Scale

Exclusion Criteria:

* Comorbid rheumatic disease (e.g., juvenile arthritis, systemic lupus erythematous)
* untreated major psychiatric diagnoses (e.g., major depression, bipolar disorder, psychoses)
* documented developmental delay
* any medical condition determined by their physician to be a contraindication for participation
* on stable medications for 4 weeks prior to enrollment
* currently in CBT or structured physical therapy program

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susmita Kashikar-Zuck, PhD, Principal Investigator — Cincinati Children's Hospital Medical Center
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fibromyalgia Integrative Training | Cognitive Behavioral Therapy
Started | 20 | 20
Post-treatment | 17 | 19
Completed | 17 | 19
Not Completed | 3 | 1
Not completed — Parent illness | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibromyalgia Integrative Training | Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.15 (1.69) | 15.50 (1.36) | 15.33 (1.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 18 | 37
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Intensity
Description: Average pain intensity in the past week marked on a paper-pencil Visual Analog Scale (Min = 0 {no pain} to Max = 10 {pain as bad as it can be}). Lower scores mean better outcomes.
Time Frame: Baseline, post-treatment and 3-month follow-up
Population: 20 participants randomized in each group. 3 dropped out of study before post-treatment and follow-up assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibromyalgia Integrative Training | Cognitive Behavioral Therapy
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 6.26 (2.06) | 6.41 (1.59)
  Post-treatment: number analyzed (Participants) | 17 | 19
  Post-treatment | 4.69 (2.13) | 6.38 (2.31)
  Primary endpoint (3-month f/u): number analyzed (Participants) | 17 | 19
  Primary endpoint (3-month f/u) | 4.62 (1.90) | 6.55 (1.22)
Statistical Analysis 1: Comparison: Fibromyalgia Integrative Training vs Cognitive Behavioral Therapy; This analysis represents the between group comparisons (i.e., FIT Teens vs. CBT) from baseline assessment to the 3-month follow-up, the primary endpoint of the trial; Test type: Superiority; p = .011, ANCOVA — The a priori threshold was alpha = .05; Adjusted for age and baseline pain levels

2. Secondary Outcome: Functional Disability
Description: Validated 15-item patient-report measure of difficulties in physical, social and recreational activities in the past 2 weeks (score Min = 0, Max = 60; Lower score means less disability/better outcome)
Time Frame: Baseline, post-treatment and 3-month follow-up
Population: 20 participants randomized to each group. 4 participants dropped out prior to post-treatment and follow-up assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibromyalgia Integrative Training | Cognitive Behavioral Therapy
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 26.70 (7.27) | 24.45 (8.29)
  Post-treatment: number analyzed (Participants) | 17 | 19
  Post-treatment | 18.71 (4.61) | 23.95 (11.04)
  Primary endpoint (3 month f/u): number analyzed (Participants) | 17 | 19
  Primary endpoint (3 month f/u) | 19.76 (5.55) | 22.68 (9.01)
Statistical Analysis 1: Comparison: Fibromyalgia Integrative Training vs Cognitive Behavioral Therapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .055, ANCOVA — The a priori threshold was alpha = .05; Adjusted for age and baseline pain levels

3. Secondary Outcome: Depressive Symptoms
Description: Children's Depression Inventory: a 27-item validated patient-report measure of depressive symptoms in the past 2 weeks (scores 0 = no depressive symptoms to 54 = most severe symptoms; lower score means less depression/better outcomes)
Time Frame: Baseline, Post-treatment, 3-month follow-up
Population: 20 participants randomized to each group. 4 participants dropped out prior to post-treatment and follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia Integrative Training | Cognitive Behavioral Therapy
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 15.8 (6.85) | 14.05 (6.18)
  Post-Treatment: number analyzed (Participants) | 17 | 19
  Post-Treatment | 11.71 (5.7) | 13.79 (7.56)
  3-month Follow-up: number analyzed (Participants) | 17 | 19
  3-month Follow-up | 11.35 (6.52) | 12.95 (7.55)

ADVERSE EVENTS:
Time Frame: Five months (2 months in active treatment and 3 month follow-up phase)
Description: The interventions in this study were purely behavioral and did not place any participants at risk for mortality or serious adverse events.
Arm/Group | Fibromyalgia Integrative Training | Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibromyalgia Integrative Training (N=20) | Cognitive Behavioral Therapy (N=20)
Joint pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Accidental injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — sports injury
Pseudo-neurologic symptoms (Psychiatric disorders) | 2 (2) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No